CLINICAL TRIAL: NCT06445504
Title: A Prospective, Multi-center, Single-arm Study of the Medtronic Hugo™ Robotic Assisted Surgery (RAS) System in Inguinal and Ventral Hernia Repair Surgery (Enable Hernia)
Brief Title: Medtronic Hugo™ Robotic Assisted Surgery (RAS) System in Hernia Surgery (Enable Hernia Repair)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT21022
Record Dates: First submitted 2024-04-01; First posted 2024-06-06 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Inguinal Hernia; Ventral Hernia
MeSH Terms: conditions — Hernia, Inguinal; Hernia, Ventral | interventions — Robotic Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Robotic-Assisted Surgery (RAS) Hernia Repair Surgery (Experimental): Patients indicated for Robotic-Assisted Surgery (RAS) for ventral and inguinal hernia repair will have the RAS surgery using the Medtronic Hugo RAS system
  Interventions: Device: Robotic-Assisted Surgery (RAS) Hernia Repair Surgery

INTERVENTIONS:
Device: Robotic-Assisted Surgery (RAS) Hernia Repair Surgery — Patients indicated for Robotic-Assisted Surgery (RAS) for ventral and inguinal hernia repair will have the RAS surgery using the Medtronic Hugo RAS system

SUMMARY:
A prospective, multicenter, single-arm pivotal study will be performed with 192 subjects enrolled to have an inguinal or ventral robotic hernia repair procedure using the Medtronic Hugo™ RAS system. Subjects will be followed through two years. This study will be conducted using up to ten investigative sites in the United States (US).

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (age ≥ 22 years) as required by local law
* Subject has been indicated for one of the following hernia repairs: (a.) primary or incisional ventral hernia(s). Multiple small hernia defects are allowed with total distance of combined defects being < 10cm (b.) inguinal (unilateral or bilateral) hernia(s).
* Subject is an acceptable candidate for a fully robotic assisted surgical procedure, a laparoscopic surgical procedure, or an open surgical procedure
* The subject is willing to participate and consents to participate, as documented by a signed and dated informed consent form

Exclusion Criteria:

* Patients for which minimally invasive surgery is contraindicated as determined by the Investigator
* Patients with a recurrent hernia
* Subjects with femoral hernia defects
* Subjects with ventral hernia defect(s) located in M1, M5, or L4
* Patients with emergent hernia repair
* Ventral hernia is CDC (Center for Disease Control) grade 2 or higher
* Use of component separation techniques to close the hernia defect
* Inability to close the hernia defect
* Hernia defect is ≥ 10 cm
* Patient has BMI > 40
* Patients with comorbidities or medical characteristics, which would preclude the surgical procedure in the opinion of the Investigator
* Patients diagnosed with a bleeding disorder and/or cannot be removed from their anticoagulants prior to surgery based on surgeon discretion and standard-of-care
* Female patients pregnant at the time of the surgical procedure.
* Patients who are considered to be part of a vulnerable population (e.g., prisoners or those without sufficient mental capacity)
* Patients who have participated in an investigational drug or device research study within 30 days of enrollment that would interfere with this study
* Patients with active infections including but not limited to pneumonia, urinary tract infection, cellulitis, or bacteremia

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2024-04-08 (Actual); Primary Completion 2025-03-19 (Actual); Study Completion 2027-03-15 (Estimated)

PRIMARY OUTCOMES:
Surgical success rate | 2 Years
  Rate of conversions from Hugo™ System to laparoscopic, open surgery, or use of an alternative robotic-assisted system.
Surgical site event rate | 2 Years
  The primary safety endpoint is the overall rate of subjects with one or more procedure- and/or device-related surgical site events (SSEs), from the first incision through 30 days post-procedure. SSE is defined as the following complications:
  * Surgical-site occurrence (SSO): Bleeding, Hemorrhage: Requiring transfusion; Bowel Injury; Bowel Obstruction; Cellulitis; Epigastric Vessel Injury; Symptomatic Hematoma: Requiring procedural intervention; Symptomatic Seroma: Requiring procedural intervention; Symptomatic Edema: Requiring procedural intervention
  * Surgical-site infection (SSI): Infection occurring where the surgery took place, including superficial, deep, and organ space infections (standardized definition developed by the CDC)

SECONDARY OUTCOMES:
Complication rate | 30 Days
  Overall rate of patients with one or more complications (Clavien-Dindo Grade I or higher), from the first incision through 30 days post-procedure.
Operative time | Intraoperative
  Time from skin incision to skin closure.
Major Complication Rate | 30 Days
  Overall rate of subjects with one or more major procedure- and/or device-related complications (Clavien-Dindo Grade III or higher), from the first incision through 30 days post-procedure.
Readmission rate through 30 days post-procedure | 30 Days
  Admission for a direct consequence or complication associated with the treated hernia or with the surgical procedure to treat the hernia.
Reoperation rate through 30 days post-procedure | 30 Days
  Operation for a direct consequence or complication associated with the treated hernia or with the surgical procedure to treat the hernia.
Recurrence rate through 2 years post-procedure | 2 Years
  Clinical hernia recurrence is defined as a palpable fascial defect and/or a clinically manifested bulge within 7 cm of the original repair, exacerbated by a Valsalva maneuver during physical examination by a study investigator. Suspected hernia recurrence(s) reported by a subject, but not confirmed by an investigator, will not be considered as a clinical hernia recurrence for this endpoint, but will be reported separately as a subject-reported recurrence.
Recurrence rate through 30 days post-procedure | 30 Days
  Clinical hernia recurrence is defined as a palpable fascial defect and/or a clinically manifested bulge within 7 cm of the original repair, exacerbated by a Valsalva maneuver during physical examination by a study investigator.

OTHER OUTCOMES:
Adverse Events (AEs) | 2 Years
  Device- and/or procedure-related AEs through 2 years.
Hospital length of stay | 30 Days
  Hospital length of stay.
Mortality rate | 30 Days
  All cause mortality.
Surgeon experience | 30 Days
  Surgeon experience survey collected after the first procedure and after the tenth procedure. If the surgeon conducts fewer than ten procedures in the study, the second survey will be conducted after the final procedure.
Pain scores | 3 Months
  Collecting ACHQC questionnaire (numerical scale where the higher the score, the greater the pain) at baseline, 30 days, and 3 months.
Transfusion rate | 30 Days
  Transfusion rate through 30 days.
Blood loss | Intraoperative
  Estimated intraoperative blood loss.
Readmission rate through 2 years | 2 Years
  Admission for a direct consequence or complication associated with the treated hernia or with the surgical procedure to treat the hernia.
Reoperation rate through 2 years | 2 Years
  Operation for a direct consequence or complication associated with the treated hernia or with the surgical procedure to treat the hernia.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Greenberg, MD, Principal Investigator — Duke University
Locations (7):
- United States (7):
  - Tampa General Hospital, Tampa, Florida
  - University of Illinois, Chicago, Chicago, Illinois
  - University of Buffalo, Buffalo, New York
  - Duke University, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - UT Health, Houston, Texas
  - Bon Secours, Newport News, Virginia

IPD SHARING:
Plan to Share IPD: Undecided